CLINICAL TRIAL: NCT00617955
Title: Systemic Effects of Aprotinin During Cardiac Surgery/ Long Term Death Rates
Brief Title: Effects of Aprotinin During Cardiac Surgery/Long Term Death Rates
Status: Completed | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Nancy A. Nussmeier, MD, SUNY Upstate Medical University, Dept. of Anesthesiology
Other Study IDs: Aprotinin; IRB Exempt #10-06; IRB #5571; NDI Y7-X070
Record Dates: First submitted 2008-02-06; First posted 2008-02-18 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2009-12

CONDITIONS: Cardiac Surgery
MeSH Terms: interventions — Aprotinin; Aminocaproic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Surgical: Cardiac surgery patients that received Aprotinin or Amicar
  Interventions: Drug: Aprotinin; Drug: Amicar

INTERVENTIONS:
Drug: Aprotinin — compare outcomes of Aprotinin versus Amicar
Drug: Amicar — compare outcomes of Aprotinin versus Amicar

SUMMARY:
The dept. of Anesthesiology currently has a database of subjects whom had surgery and received either Aprotinin or Amicar in the OR. The current viewpoint is that Aprotinin is more harmful than Amicard. In an effort to see what the long term outcomes were for subjects whom had surgery here at Upstate, it was decided to look at long term death rates to see if any differences. A student t-test will be used to determine statistical significance where a p value of <0.05 will be deemed significant. Using data from 462 subjects that had undergone cardiac surgery at SUNY Upstate Medical University, CABG only and the long term mortality rate from the Mangano, et.al. publications, the unadjusted mortality for the two drugs are Aprotinin 5.4% and Amicar 1.2%. A power analysis was performed using the hospital mortality rates of 5.4% and 1.2% with the sample size in the propensity data and a p-value of 0.05. The result was a power of 81.7%.

DETAILED DESCRIPTION:
Charts for 462 subjects will be reviewed from 2002-2005 based on the surgery performed. From each chart, the subject name, date of birth,and social security number will be recorded along with the state of residence and year of surgery. This information will be transferred to a CD that is encrypted and password protected. The CD will be sent via FedEx overnight to the Center for Disease Control(CDC), National Death Registry. The CDC will use the information on the CD to extract death outcomes for each subject's information provided. Once all information is complete, the CDC will transfer on to a CD that is encrypted and password protected and return to our office via FexEx overnight. The information on the CD will then be used to determine what the long term death rates were for subjects here at SUNY Upstate Medical University and stored in an anonymous database. Once the information is verified as accurate, the CD will be destroyed and no identifying information will be kept. The CDC will also destroy the information after 60 days, with no links to the identifying information.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 years of age or older
* Subjects must have received either Aprotinin or Amicar during cardiac surgery

Exclusion Criteria:

* Cardiac surgery and did not receive Aprotinin or Amicar

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiac Surgery patients
Sampling Method: Probability Sample
Enrollment: 462 (Actual)
Dates: Start 2007-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Long term death rates | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Nancy A Nussmeier, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States